CLINICAL TRIAL: NCT05163873
Title: ExPECT: Extraperitoneal End Colostomy Trial - Feasibility Phase
Brief Title: ExPECT: Extraperitoneal End Colostomy Trial
Acronym: ExPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea Bay University Health Board (Other)
Collaborators: Swansea University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 291897
Record Dates: First submitted 2021-11-08; First posted 2021-12-20 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Colostomy Stoma; Cancer of Colon; Surgery; Quality of Life
Keywords: colostomy; surgery; colon cancer; feasibility study; cancer
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans-peritoneal (No Intervention): Surgery technique in the formation of permanent end colostomy
- Extra-peritoneal (Experimental): Surgery technique in the formation of permanent end colostomy
  Interventions: Procedure: Extra-peritoneal

INTERVENTIONS:
Procedure: Extra-peritoneal — Surgery procedure: a non-mesh prophylactic surgical technique to prevent PH
  Arms: Extra-peritoneal

SUMMARY:
A randomised controlled feasibility study to compare two surgery techniques in the formation of a permanent end colostomy; the trans-peritoneal(TP) technique - currently, the most commonly used technique and the investigational extra-peritoneal(EP) technique, which has been reported in small studies to reduce the risk of parastomal hernia . This feasibility study will primarily aim to determine the feasibility viability of progression to a full multi-centre trial and test study design acceptability for participants. Participants will be asked to consent to be randomised to either the TP or EP procedure during surgery. Following surgery, participants will be followed up to a maximum of 12 months and asked to complete quality of life questionnaires (EQ5D and Colostomy Impact Score). Participant data will also be accessed by research teams at site to collect data on stoma appliance use and complications.

DETAILED DESCRIPTION:
This feasibility study is a multi-centre, single (patient) blinded, randomised controlled trial (RCT). Co-ordination and trial management will be led from Swansea Trials Unit (STU).

The study will take place across 3 sites: Swansea Bay University Health Board (SBUHB); Aneurin Bevan University Health Board and Cardiff and Vale University Health Board. Surgeons at all three sites have experience with both interventional extra-peritoneal surgical technique and the most commonly used transperitoneal technique.

The investigators aim to recruit 60 participants over 12 months. Local recruitment will be co-ordinated by PIs and research teams. Recruitment is aimed to be equally distributed across all sites. Participants will be equally randomised by arm in each of the three sites: to receive the EP colostomy formation (Intervention) or the standard transperitoneal (TP) technique. Participants will remain blinded as to their treatment until the close of the study.

Data collection will be performed by the clinical and research teams, with support from PIs. Data will be stored centrally in REDCap (Research Electronic Data Capture) software.

The investigators will explore whether it is possible to establish a research infrastructure in which data can be collected and co-ordinated across sites and for patients to be followed up effectively. The investigators will also look to demonstrate standardisation of the operative technique for EP stoma formation and to determine which outcome measures a future trial should explore. This feasibility trial be evaluated against ACCEPT progression criteria.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* Able and willing to give informed consent to participate
* Elective patient for colorectal surgery requiring formation of permanent end colostomy (This may include patients undergoing surgery for rectal or anal cancer, inflammatory bowel disease, diverticular disease and functional bowel disorders)
* Suitable to receive both trans-peritoneal and extra-peritoneal techniques

Exclusion Criteria:

* Lacking the capacity to consent
* Having emergency surgery
* Previous or current abdominal wall stoma
* Intention to form loop colostomy, ileostomy or double-barrelled stoma
* Previous incisional hernia repair with disruption of abdominal wall layers
* Pregnant or breastfeeding (as determined by standard NHS procedures)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Assessing the feasibility of the trial based on recruitment rate | Consent
  number of eligible patients who consent
Assessing the feasibility of the trial based on data completeness | Week 6
  % follow up data collected for 80% of participants
Assessing the feasibility of the trial based on surgeon involvement | set up
  number of surgeons at sites willing to be involved in the trial
Assessing the feasibility of the trial based on recruitment within sites | consent
  number of patients recruited at each site to be at least 10
Assessing the feasibility of the trial based on surgeon training | set up
  ability to successfully train surgeons taking part
Assessing the feasibility of the trial based on surgeon compliance with the intervention | month 12
  80% compliance with the correct technique required
Assessing the feasibility of the trial based on collection of key outcomes | week 6, month 6 and month 12
  collection of colostomy impact score, EQ-5D and rate of parastomal hernia
Assessing the feasibility of the trial based on overall QoL reported in intervention group compared with standard care group | week 6, month 6 and month 12
  QoL data to be 80% or more of that in the standard care group

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Taylor, Study Director — Swansea Bay University Health Board
Locations (3):
- United Kingdom (3):
  - Cardiff and Vale University Health Board, Cardiff
  - Aneurin Bevan University Health Board, Newport
  - Swansea Bay University Health Board, Swansea

IPD SHARING:
Plan to Share IPD: No
No current plan to share IPD but will discuss with study team if and/or when the request arises.